CLINICAL TRIAL: NCT04602910
Title: Developing a Web-based Shared Decision-making Tool for Fertility Preservation Among Reproductive-age Women With Breast Cancer: An Action Research Approach
Brief Title: Developing a Web-based Shared Decision-making Tool for Fertility Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chin-Tsung Shen, Mackay Medical College, Mackay Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSM/VGH-V108E-005-1
Record Dates: First submitted 2020-10-15; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Breast Neoplasm Female
Keywords: breast cancer; shared decision making; website; action research; fertility preservation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the phases of planning and acting (Experimental): Each part of the website page was assessed for comprehensibility and usability by patients. Health care providers were asked to assess the acceptability of the website. A 5-point Likert scale was used for patient and health care provider ratings for each item. If the score were less than 3, then we would modify the website content based on the user feedback from patients and health care providers
  Interventions: Device: a web-based shared decision-making tool

INTERVENTIONS:
Device: a web-based shared decision-making tool — Five major parts were developed with the use of the action research approach. The Introduction and Options (parts 1 and 2) describe the severity of the cancer treatment and infertility and the knowledge of fertility preservation, respectively. The SDM tool was designed as a step by step process (part 3) that involves the comparison of options, patient's values and preferences, their knowledge regarding infertility and options, and reaching a collective decision. The Resources (part 4) provide information on the hospitals that provide such services, and the References (part 5) list all the literature cited in the website. The results show the web-based SDM meets both the patients' and health providers' needs and helps reproductive-age patients with breast cancer make decisions on fertility preservation.

SUMMARY:
The objective of this study was to develop a web-based, shared decision-making (SDM) tool for helping patients with breast cancer make decisions on fertility preservation.

DETAILED DESCRIPTION:
Background: The pregnancy rate after cancer treatment for female survivors is lower than that of the general population. Future infertility is a significant concern for patients with breast cancer and is associated with a poor quality of life. Reproductive- age patients with breast cancer have safe options when choosing the type of fertility preservation method to be applied. Better information and support resources aimed at women to support their decision making are needed.

Objective: The objective of this study was to develop a web-based, shared decision-making (SDM) tool for helping patients with breast cancer make decisions on fertility preservation.

Methods: We used the action research cycle of observing, reflecting, planning, and acting to develop a web-based SDM tool. The following four phrases were applied: (1) Observe and reflect: Collect and analyze the decision-making experiences of patients and health care providers; (2) Reflect and plan: Apply the initial results to create a paper design and modify the content; (3) Plan and act: Brainstorm about the web pages, and modify the content; (4) Act and observe: Evaluate the effectiveness, and refine the website SDM. Interviews, group meetings, and constant dialogue were conducted between the various participants at each step. The effectiveness was evaluated using the Preparation for Decision-Making (prepDM) scale.

ELIGIBILITY:
Inclusion Criteria:

* Health provider who ever cared the patients with breast cancer.
* Patients with breast cancer who are younger than 50 years old.

Exclusion Criteria:

* none

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Preparation for Decision-Making | 1 week
  We evaluated the effectiveness of the Preparation for Decision-Making (prepDM) scale. Both patients and health care providers were invited to answer 10 questions by responding with a 5-point Likert scale rating (from 1 to 5). A higher score indicated greater agree with the effect.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Miauh Huang, PhD, Principal Investigator — Department of Nursing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng LM, Lien PJ, Huang CY, Tsai YF, Chao TC, Huang SM. Developing a Web-Based Shared Decision-Making Tool for Fertility Preservation Among Reproductive-Age Women With Breast Cancer: An Action Research Approach. J Med Internet Res. 2021 Mar 17;23(3):e24926. doi: 10.2196/24926. PMID 33729164
- See also: a web-based shared decision-making tool for fertility preservation among reproductive-age women with breast cancer — http://vghtpe-cbhc.sdmcare.me/healthEducation